CLINICAL TRIAL: NCT03416166
Title: International Multisite Transcatheter Tricuspid Valve Therapies Registry
Acronym: TriValve
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-01753
Record Dates: First submitted 2018-01-23; First posted 2018-01-30 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Severe Tricuspid Regurgitation
Keywords: Tricuspid Valve; tricuspid regurgitation; transcatheter tricuspid regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Transcatheter Tricuspid Intervention — Any available transcatheter tricuspid valve intervention

SUMMARY:
For a long time, tricuspid valve disease has been considered as less important than left-sided valvular heart disease. If treated in an advanced stage and simultaneously with other cardiac diseases, it is associated with significant morbidity and mortality. Hence, physicians tend to refer patients more aggressively to surgery (1).

Transcatheter procedures are an attractive alternative in high-risk patients. The field of transcatheter tricuspid devices has rapidly advanced over the last few years (2). Limited knowledge is available regarding the epidemiologic and anatomical settings in which these therapies are preferentially applied.

The main purpose of this registry is the collection of baseline clinical and anatomical data of the patients treated with transcatheter tricuspid valve therapies, and their outcomes, whenever feasible. Apart from more knowledge regarding the current status in this field, the results could also help the establishment of guidelines with respect to the choice of the transcatheter device selected and to understand which therapy can provide the better outcome in the different anatomies. Moreover, this study will provide important information about the epidemiology of severe tricuspid regurgitation, which is at the moment an undertreated disease.

ELIGIBILITY:
Inclusion Criteria:

* All the patients undergoing transcatheter tricuspid valve intervention.

General inclusion criteria:

* Minimal age: 18 years
* Patient is able to give written informed consent to the procedure

Exclusion Criteria:

* Patients not fulfilling the indications for transcatheter tricuspid intervention

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with severe symptomatic tricuspid regurgitation
Sampling Method: Non-Probability Sample
Enrollment: 269 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular Death | 30 days

SECONDARY OUTCOMES:
NYHA Class | 30 days, 1 year
TR Reduction | 30 days, 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Scotti A, Coisne A, Taramasso M, Granada JF, Ludwig S, Rodes-Cabau J, Lurz P, Hausleiter J, Fam N, Kodali SK, Rosiene J, Feinberg A, Pozzoli A, Alessandrini H, Biasco L, Brochet E, Denti P, Estevez-Loureiro R, Frerker C, Ho EC, Monivas V, Nickenig G, Praz F, Puri R, Sievert H, Tang GHL, Andreas M, Von Bardeleben RS, Rommel KP, Muntane-Carol G, Gavazzoni M, Braun D, Koell B, Kalbacher D, Connelly KA, Juliard JM, Harr C, Pedrazzini G, Russo G, Philippon F, Schofer J, Thiele H, Unterhuber M, Himbert D, Alcazar MU, Wild MG, Windecker S, Jorde U, Maisano F, Leon MB, Hahn RT, Latib A. Sex-related characteristics and short-term outcomes of patients undergoing transcatheter tricuspid valve intervention for tricuspid regurgitation. Eur Heart J. 2023 Mar 7;44(10):822-832. doi: 10.1093/eurheartj/ehac735. PMID 36445158
- [Derived] Muntane-Carol G, Taramasso M, Miura M, Gavazzoni M, Pozzoli A, Alessandrini H, Latib A, Attinger-Toller A, Biasco L, Braun D, Brochet E, Connelly KA, de Bruijn S, Denti P, Deuschl F, Lubos E, Ludwig S, Kalbacher D, Estevez-Loureiro R, Fam N, Frerker C, Ho E, Juliard JM, Kaple R, Kodali S, Kreidel F, Harr C, Lauten A, Lurz J, Monivas V, Mehr M, Nazif T, Nickening G, Pedrazzini G, Philippon F, Praz F, Puri R, Schafer U, Schofer J, Sievert H, Tang GHL, Khattab AA, Andreas M, Russo M, Thiele H, Unterhuber M, Himbert D, Urena M, von Bardeleben RS, Webb JG, Weber M, Windecker S, Winkel M, Zuber M, Hausleiter J, Lurz P, Maisano F, Leon MB, Hahn RT, Rodes-Cabau J. Transcatheter Tricuspid Valve Intervention in Patients With Right Ventricular Dysfunction or Pulmonary Hypertension: Insights From the TriValve Registry. Circ Cardiovasc Interv. 2021 Feb;14(2):e009685. doi: 10.1161/CIRCINTERVENTIONS.120.009685. Epub 2021 Feb 5. PMID 33541097
- [Derived] Miura M, Alessandrini H, Alkhodair A, Attinger-Toller A, Biasco L, Lurz P, Braun D, Brochet E, Connelly KA, de Bruijn S, Denti P, Deuschl F, Estevez-Loureiro R, Fam N, Frerker C, Gavazzoni M, Hausleiter J, Himbert D, Ho E, Juliard JM, Kaple R, Besler C, Kodali S, Kreidel F, Kuck KH, Latib A, Lauten A, Monivas V, Mehr M, Muntane-Carol G, Nazif T, Nickenig G, Pedrazzini G, Philippon F, Pozzoli A, Praz F, Puri R, Rodes-Cabau J, Schafer U, Schofer J, Sievert H, Tang GHL, Thiele H, Rommel KP, Vahanian A, Von Bardeleben RS, Webb JG, Weber M, Windecker S, Winkel M, Zuber M, Leon MB, Maisano F, Hahn RT, Taramasso M; TriValve Investigators. Impact of Massive or Torrential Tricuspid Regurgitation in Patients Undergoing Transcatheter Tricuspid Valve Intervention. JACC Cardiovasc Interv. 2020 Sep 14;13(17):1999-2009. doi: 10.1016/j.jcin.2020.05.011. PMID 32912460